CLINICAL TRIAL: NCT05163457
Title: Prevalence of Frailty Among People Aged 75 and Over Living at Home
Acronym: FRAIL-DOM
Status: Completed | Type: Observational
Sponsor: Université de Reims Champagne-Ardenne (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-012-FRAIL-DOM
Record Dates: First submitted 2021-12-06; First posted 2021-12-20 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2022-03

CONDITIONS: Frailty
Keywords: Frailty - SEGAm - living at home
MeSH Terms: conditions — Frailty | interventions — Data Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- aged of 75 and more living at home: aged of 75 and more living at home" group: patients aged of 75 and more living at home
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection — frailty evaluation

SUMMARY:
The aging of population lead to study ways to prevent dependence. Frailty is a precursor to dependence which can be reversible. In the literature, estimate of prevalence of frailty is highly variable depending on the frailty definition, the population studied and the screan tool used. In fact, many scales to measure frailty have emerged without gold standard.

The SEGAm showed its usefulness in aged patients living at home.

DETAILED DESCRIPTION:
The aim of the study is to describe prevalence of frailty in patients aged of 75 and more living at home.

ELIGIBILITY:
Inclusion Criteria:

* male or female
* aged of 75 and more
* living at home
* agreeing to participate in the study

Exclusion Criteria:

- none

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: patients aged of 75 and more living at home
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2022-01-06 (Actual); Primary Completion 2022-02-22 (Actual); Study Completion 2022-02-22 (Actual)

PRIMARY OUTCOMES:
Frailty | Day 0
  Frailty evaluated using SEGA modified scale (SEGAm). SEGAm includes 13 items (coded from 0 to 2) to obtain a global score out of 26 points. Patients with a score less than or equal to 8 are considered not fragile. Patients with a score between 8 and 11 are considered fragile. Patients with a score greater than or equal to 11 are considered very fragile.

CONTACTS AND LOCATIONS:
Locations (1):
- Maison de Santé Pluridisciplinaire de Bar sur Seine, Bar-sur-Seine, Grand Est, France

IPD SHARING:
Plan to Share IPD: No